CLINICAL TRIAL: NCT01175161
Title: A Pilot Study Of A Randomized Trial Comparing Two Different Time Frames For Copper T380A Intrauterine Contraception Insertion; Immediately Postpartum Compared To 4-6 Weeks Postpartum In Lilongwe, Malawi
Brief Title: Postpartum Intrauterine Device Study
Acronym: PPIUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Amy Bryant, Fellow, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CID-0925
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Contraception; Intrauterine Devices; Pilot Study; Africa
Keywords: Postpartum Contraception; Intrauterine device; feasibility; IUD; Immediate postpartum IUD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate postpartum IUD insertion (Experimental): Women assigned to have the IUD placed 10 minutes to 48 hours postpartum
  Interventions: Device: Copper T380A Intrauterine Device
- 6 week postpartum IUD insertion (Experimental): Women who receive the IUD at the traditional time frame.
  Interventions: Device: Copper T380A Intrauterine Device

INTERVENTIONS:
Device: Copper T380A Intrauterine Device — the Copper T380A IUD will be placed either 10 minutes to 48 hours postpartum, or 4-6 weeks postpartum.

SUMMARY:
The purpose of this non-blinded randomized clinical trial is to pilot the design of a randomized clinical trial to be conducted in Malawi to investigate immediate postpartum insertion of the Copper T380 intrauterine contraceptive device (CuT380A-IUCD) compared to placement at the 6-week postpartum visit.

The investigators hypothesize that it will be feasible to enroll 140 women into this study, and that women will find the 10 minute to 48 hour time frame for IUCD placement acceptable.

DETAILED DESCRIPTION:
Women will be enrolled into the study during prenatal care. After delivery, if they meet secondary eligibility criteria, they will be randomized to receive the IUD immediately postpartum or at the 6-week postpartum visit. Women will be followed at 4, 8, and 12 weeks after IUD insertion, and be assessed at those time points for satisfaction with the method and IUD expulsion.

ELIGIBILITY:
Inclusion Criteria:

* Primary Inclusion Criteria:

  * Ages 18-45 attending prenatal care
  * Greater than 34 weeks estimated gestational age
  * Desire to use the CuT380A-IUCD for contraception postpartum
  * Plan to stay in the area for at least 5 months postpartum
  * If HIV+ the women must be WHO Clinical Stage 1 or 2, or known to be clinically well on antiretroviral therapy as documented in their health passport
  * No prior cesarean delivery
  * No treatment for pelvic inflammatory disease within 3 months prior to pregnancy
  * No known uterine anomalies
  * No known pelvic tuberculosis
  * No known genital tract cancer
  * No known allergy to copper
  * No known history of ectopic pregnancy within 3 months prior to pregnancy.
  * No evidence of clinical anemia as assessed by a clinician at enrollment
  * Any other condition a clinician feels should preclude the woman from receiving the IUCD 10-minutes to 48 hours after delivery

Secondary Eligibility Criteria

* Vaginal delivery within the last 48 hours
* No postpartum hemorrhage documented by the delivering clinician
* Not known to have ruptured membranes for greater than 24 hours prior to delivery
* No infection diagnosed by a clinician
* No fever of greater than 38° during labour or delivery
* Any other condition which a clinician feels precludes the woman from receiving the IUCD 10 minutes to 48 hours after delivery.

Exclusion Criteria:

* prior cesarean section
* fever during labor and delivery
* AIDS, not well on antiretroviral therapy
* genital tuberculosis
* known uterine abnormalities or genital tract cancer
* history of ectopic pregnancy within 3 months of current pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Time | 6 months
  Estimate the time required to enroll 140 women into this study

SECONDARY OUTCOMES:
Expulsion rates | 6 months
  Estimate the expulsion rate of the CuT380A-IUCD
Satisfaction | 6 months
  Assess patient and provider satisfaction when the CuT380A-IUCD is placed 10 minutes - 48-hours postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Amy G Bryant, MD, Principal Investigator — University of North Carolina, Chapel Hill; Gretchen S Stuart, MD, MPHTM, Study Director — University of Carolina Chapel Hill
Locations (1):
- University of North Carolina Project Lilongwe, Lilongwe, Malawi

REFERENCES:
- [Derived] Bryant AG, Kamanga G, Stuart GS, Haddad LB, Meguid T, Mhango C. Immediate postpartum versus 6-week postpartum intrauterine device insertion: a feasibility study of a randomized controlled trial. Afr J Reprod Health. 2013 Jun;17(2):72-9. PMID 24069753